CLINICAL TRIAL: NCT00593229
Title: An Observational Study of All Forms of Thrombotic Microangiopathy in Pediatric Patients
Brief Title: International Registry and Biorepository for TMA(Thrombotic Microangiopathy)
Status: Terminated | Type: Observational
Why Stopped: study stopped at this site, as investigator left the institution
Sponsor: Northwell Health (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Mario Negri Institute for Pharmacological Research (Other); Icahn School of Medicine at Mount Sinai (Other); University of Virginia (Other); Montreal Children's Hospital of the MUHC (Other); University of Utah (Other); Stollery Children's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK71221; DK R21-71221
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Thrombotic Microangiopathy; Hemolytic Uremic Syndrome; Thrombotic Thrombocytopenic Purpura
Keywords: Thrombotic microangiopathy (TMA); Hemolytic uremic syndrome (HUS); Thrombotic thrombocytopenic purpura (TTP)
MeSH Terms: conditions — Thrombotic Microangiopathies; Hemolytic-Uremic Syndrome; Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 3: Familial atypical HUS
- 4: Thrombotic thrombocytopenic purpura (TTP)
- 1: Severe diarrhea-associated hemolytic uremic syndrome (D+HUS)
- 2: Non-familial atypical HUS

SUMMARY:
This registry will collect clinical data and store biosamples (seru, plasma, urine, and DNA) annually from pediatric patients with thrombotic mcroangiopathy

DETAILED DESCRIPTION:
Children age, 6 months - 18 years, are eligible if they have one of the following categories of thrombotic microangiopathy (TMA):(1) severe D+HUS; (2) non-familial atypical HUS; (3) familial atypical HUS; or (4) TTP

Patients are seen intially and annually thereafter

Biosamples are collected for storage annually.

ELIGIBILITY:
Inclusion Criteria:

* Severe HUS, familial or non-familial atypical HUS, TTP

Exclusion Criteria:

* None

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients, 6 months - 18 years
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Determine epidemiology and outcomes of the various forms of TMA | Ongoing
Determine genetic causes of TMA | Ongoing

SECONDARY OUTCOMES:
Initiate clinical trials in TMA | In the future

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — Schneider Children's Hospital
Locations (1):
- Schneider Chldren's Hospital, New Hyde Park, New York, United States